CLINICAL TRIAL: NCT04146506
Title: The Effect of Stretching on Pain Sensitivity - Potential Gender Differences?
Brief Title: Gender Differences in the Tolerance to Stretch
Status: Completed | Type: Observational
Sponsor: University College of Northern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: UniversityCND2
Record Dates: First submitted 2019-10-24; First posted 2019-10-31 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2019-10

CONDITIONS: Range of Motion, Articular; Muscle Stretching Exercises
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male: Static Muscle stretching exercises of the knee flexors
  Interventions: Other: Muscle stretching exercises
- Female: Static Muscle stretching exercises of the knee flexors
  Interventions: Other: Muscle stretching exercises

INTERVENTIONS:
Other: Muscle stretching exercises — Muscle stretching exercises consisting of static stretching exercises of the knee flexors

SUMMARY:
The effect of stretching on range of motion is believed to rely upon an increased tolerance to stretch. This suggests, that pain modulation has significance in regards to the effect of stretching.

DETAILED DESCRIPTION:
Given that there may be differences in the way men and women perceive a painful stimulus, this suggests that there may be potential gender differences in the tolerance to stretch following stretching.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any pain or other conditions which might affect the somatosensory system and pain perception

Exclusion Criteria:

* Substance abuse, History of neurological or mental disabilities, Lack of ability to comply with instructions, Delayed onset of muscle soreness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female volunteers between the ages of 18 to 45 are eligible for participation.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Range of Motion | Passive knee extension range of motion was measured at baseline just prior to Muscle stretching exercises
  Passive knee extension Range of motion
Range of Motion | Passive knee extension range of motion was measured 30 seconds after Muscle stretching exercises
  Passive knee extension Range of motion
Pain Thresholds | Pressure pain Thresholds were measured at baseline just prior to muscle stretching exercises
  Pressure Pain Thresholds
Pain Thresholds | Pressure pain Thresholds were measured 30 seconds after muscle stretching exercises
  Pressure Pain Thresholds
Torque | Passive resistive torque was measured at baseline just prior to muscle stretching exercises
  Passive Resistive Torque
Torque | Passive resistive torque was measured 30 seconds after muscle stretching exercises
  Passive Resistive Torque

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Drachman, Msc., Study Director — University College of Northern Denmark, Department of Physiotherapy
Locations (1):
- University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD (range of motion, PPT and Torque data) will be shared upon request